CLINICAL TRIAL: NCT00595933
Title: A Comparative Trial of Over-the-counter Dry Mouth Remedies for Dry Mouth After Radiation to the Head and Neck
Brief Title: Comparing Over-the-counter Dry Mouth Remedies After Radiation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Dry Mouth_Krempl; IRB # 12518 (Other: Institutional Review Board)
Record Dates: First submitted 2007-12-20; First posted 2008-01-16 (Estimated); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Xerostomia
Keywords: Head and Neck cancer; Radiation therapy; Dry mouth remedies; Dry Mouth; Xerostomia
MeSH Terms: conditions — Xerostomia; Head and Neck Neoplasms | interventions — Chewing Gum; Mouthwashes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Each participant will receive an unidentified product to use for a one week period. This will continue until all 7 dry-mouth products have been evaluated.
  Interventions: Other: sugar-free chewing gum; Other: chewing gum; Other: mouth rinse; Drug: mouth spray

INTERVENTIONS:
Other: sugar-free chewing gum — Chew gum 4 times a day with additional allowances for as needed. Fill out daily questionaire and an end of week.
  Other Names: Freedent chewing gum
Other: chewing gum — Chew gum 4 times a day with additional allowances for as needed. Fill out daily questionaire and an end of week.
  Other Names: Biotene chewing gum
Other: mouth rinse — Rinse mouth 4 times a day with additional allowances for as needed. Fill out daily questionaire and an end of week questionaire
  Other Names: Flavored water
Other: mouth rinse — Rinse mouth 4 times a day with additional allowances for as needed. Fill out daily questionaire and an end of week.
  Other Names: Biotene mouth rinse
Drug: mouth spray — Spray mouth with mouth spray 4 times a day with additional allowances for as needed. Fill out daily questionaire and an end of week
  Other Names: Salivart
Drug: mouth spray — Spray mouth 4 times a day with additional allowances for as needed. Fill out daily questionaire and an end of week
  Other Names: MouthKote

SUMMARY:
The purpose of this study is to compare the effectiveness of over-the-counter remedies for dry mouth.

DETAILED DESCRIPTION:
Xerostomia (dry mouth) is the most common late complication of radiation therapy for head and neck cancers. When patients are cured or survive for several years, xerostomia often becomes quite bothersome; it affects their quality of life. This study compares the effectiveness of seven over-the-counter remedies, 2 rinses, 3 sprays and 2 chewing gums. A computer program will make random assignments so that the patient nor the physician will choose the order in which the products are tried. The remedies will be used for one week each and at the end of each period the patient will fill out a questionaire.

ELIGIBILITY:
Inclusion Criteria:

* Suffers from Xerostomia
* Surviver of head and neck cancer that received >5000 cGy radiation therapy >1 year prior to study entry.
* Able to chew, rinse and swallow.
* Ages 13-99 years of age

Exclusion Criteria:

* Currently using the following medications: anorexiants, antiacne agents, Anticholinergic agents, tricyclic antidepressants, chemotherapy agents.
* Unable to complete questionnaires

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2005-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The effectiveness of seven over-the-counter remedies for dry mouth as determined by amount of saliva output and a brief questionaire. | 8-10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Greg Krempl, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States